CLINICAL TRIAL: NCT04388241
Title: Preliminary Feasibility and Efficacy of The Balance Program to Reduce the Impact of Pain on Daily Functioning in Pediatric Sickle Cell Disease
Brief Title: Preliminary Feasibility and Efficacy of Behavioral Intervention to Reduce Pain-Related Disability in Pediatric SCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Megan Connolly, PhD; Assistant Professor of Pediatrics and Psychiatry & Behavioral Sciences, Children's National Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00013663
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2022-09-06 (Actual); Status verified 2022-09

CONDITIONS: Sickle Cell Disease; Pain
MeSH Terms: conditions — Anemia, Sickle Cell; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Intervention (Experimental): Children and adolescents with SCD between the ages of 8 and 17 years old (n=20) will be recruited to complete a four-week behavioral intervention designed to reduce pain-related impairment in SCD.
  Interventions: Behavioral: The Balance Program

INTERVENTIONS:
Behavioral: The Balance Program — The Balance Program is a four-week behavioral intervention (each session lasting 60 minutes) developed specifically for the pediatric SCD population based on existing evidence-based treatments to target the unique presentation of pain-related disability in SCD.

SUMMARY:
Pain is the primary complication of sickle cell disease (SCD), including vaso-occlusive crises and more persistent, chronic pain. SCD-related pain is associated with significant functional impairment, spanning poor school attendance, decreased quality of life, and stress and mood difficulties. Pharmacological approaches are the first-line treatment for SCD-related pain, but these can be costly and have unwanted side effects. Given limitations from pharmacological approaches and the influence that poor behavioral responses have on disease management and health outcomes suggest a critical need for alternative and adjunctive treatments. Due to gaps in available behavioral treatments specifically designed for addressing common challenges associated with pain management in pediatric SCD, the investigators developed a manualized behavioral therapy protocol by tailoring existing evidence-based treatments. The overall goal of the intervention is to reduce the impact of pain on daily functioning in pediatric SCD. This study will empirically test the feasibility and preliminary efficacy of this intervention for youth with SCD. Children and adolescents with SCD between the ages of 8 and 17 years old (n=20) will be recruited to complete the treatment protocol. Feasibility will be assessed by examining participation and program completion rates, as well as feedback from a treatment acceptability questionnaire and qualitative interview. Participants will complete baseline assessments, weekly questionnaires, and post-treatment assessments (post-intervention assessment, follow-up time points: 1-month following the intervention, and 3-months following the intervention).

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with SCD (HbSS, HbSC, HbS-beta0 thalassemia, or HbS-beta+ thalassemia) between the ages of 8 and 17 years old with pain-related disability and who are currently prescribed short- or long-acting opioid medications.

  1. Participants will meet at least one of the following criteria for pain-related disability: 1) Have had at least 3 pain crises in the last year, 2) Have had at least one admission for pain in the last year, or 3) Have missed at least one week of school (5 days) in the last year
  2. Current prescription of opioids will be confirmed by participants' primary hematologist, review of the electronic medical record, and discussion with the family.

Exclusion Criteria:

* Patients and caregivers with limited English proficiency, a neurodevelopmental delay, or a visual or motor impairment that would interfere with their ability to complete the assessments and intervention.
* Documented history of major depressive disorder in medical record and/or through discussion with their primary hematology suggesting that patients may need a specific and higher level of therapeutic care.
* Patients have regularly scheduled outpatient therapy sessions outside of the study.

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2020-09-23 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-08-04 (Actual)

PRIMARY OUTCOMES:
Feasibility assessed by program completion rates | Following the completion of the intervention (5 weeks from baseline)
  Feasibility will be determined by examining the proportion of participants (e.g., 80%) that complete all four sessions.
Acceptability assessed by satisfaction ratings and report | Following the completion of the intervention (5 weeks from baseline)
  Acceptability will be determined by examining the satisfaction with the treatment on the Treatment Evaluation Inventory (TEI) (i.e., >80% reporting at least a "moderate" acceptability on the TEI) as well as through analysis of qualitative interviews.
Preliminary efficacy of the intervention in changing pain-related outcomes | Following the completion of the intervention (5 weeks from baseline, 1-month follow up, 3-month follow up))
  Efficacy will be determined by examining self- and parent-reported changes in pain-related disability and behaviors at post-intervention and one- and three- month follow-up compared to baseline
Preliminary efficacy of the intervention in changing pain-related outcomes as measured by medication use | Following the completion of the intervention (5 weeks from baseline, 1-month follow up, 3-month follow up))
  Efficacy will also be determined by examining changes in opioid use, as measured by number of prescriptions filled and self-reported use, at post-intervention and one- and three- month follow-up compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Connolly, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States